CLINICAL TRIAL: NCT00835705
Title: Randomized, 2-way Crossover, Bioequivalence Study of Amoxicillin-Clavulanic Acid 400 Mg-57 mg Chewable Tablets and AUGMENTIN® 400 Mg-57 mg Chewable Tablets Administered as 1 x 400 Mg-57 mg Chewable Tablet in Healthy Subjects Under Fasting Conditions
Brief Title: Amoxicillin-Clavulanic Acid 400 Mg-57 mg Chewable Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 30073
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amoxicillin Clavulanic Acid (Experimental): Amoxicillin Clavulanic Acid 400-57 mg Chewable Tablet (test) dosed in first period followed by Augmentin® 400-57 mg Chewable Tablet (reference) dosed in second period
  Interventions: Drug: amoxicillin-clavulanic acid
- Augmentin® (Active Comparator): Augmentin® 400-57 mg Chewable Tablet (reference) dosed in first period followed by Amoxicillin Clavulanic Acid 400-57 mg Chewable Tablet (test) dosed in second period
  Interventions: Drug: Augmentin®

INTERVENTIONS:
Drug: amoxicillin-clavulanic acid — 400 mg-57 mg chewable tablet
  Arms: Amoxicillin Clavulanic Acid
Drug: Augmentin® — 400 mg-57 mg chewable tablet
  Arms: Augmentin®

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of amoxicillin-clavulanic acid 400 mg-57 mg chewable tablets (test) versus Augmentin® (reference) administered as 1 x 400 mg-57 mg chewable tablet under fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria

* Subjects will be females and/or males, non-smokers, 18 years of age and older.

Exclusion Criteria

Subjects to whom any of the following applies will be excluded from the study:

* Clinically significant illnesses within 4 weeks of the administration of study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the medical subinvestigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive urine drug screen at screening.
* Positive testing for hepatitis B, hepatitis C or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, or diastolic blood pressure lower than 50 or over 90; or heart rate less than 50 bpm) at screening.
* Subjects with BMI ≥30.0.
* History of significant alcohol abuse within six months of the screening visit or any indication of the regular use of more than two units of alcohol per day (1 Unit = 150 mL of wine or 360 mL of beer or 45 mL of alcohol 40%).
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months of the screening visit or hard drugs (such as cocaine, phencyclidine (PCP) and crack) within 1 year of the screening visit.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the medical subinvestigator, contraindicates the subject's participation in this study.
* History of allergic or hypersensitivity reactions to amoxicillin or clavulanic acid or other related drugs (e.g. penicillin, cephalosporins, cephamycins).
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin; examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin, ketoconazole, MAO inhibitors, neuroleptics, verapamil, quinidine, valproic acid)
* use of an investigational drug or participation on an investigation study within 30 days prior to the administration of the study medication.
* Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
* Any clinically significant history or presence of clinically significant neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric or metabolic disease.
* Any food allergy, intolerance, restriction or special diet that could, in the opinion of the Medical Subinvestigator, contraindicate the subject's participation in this study.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products )including natural products, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Subjects who have had a depot injection or an implant of any drug 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days. Donation or loss of whole blood prior to administration of the study medication as follows:
* Less than 300 mL of whole blood within 30 days or
* 300 mL to 500 mL of whole blood within 45 days or
* more than 500 mL of whole blood within 56 days.
* Positive alcohol breath test at screening.
* Subjects who have used tobacco in any form within the 90 days preceding study drug administration.
* Intolerance to venipunctures
* Subjects with a clinically significant history of tuberculosis, epilepsy, asthma, diabetes, psychosis, or glaucoma will not be eligible for this study.
* Any history of known Augmentin-associated cholestatic jaundice/hepatic dysfunction
* Any known active mononucleosis
* Subjects with dentures or braces.

Additional exclusion criteria for female subjects only:

* Breast feeding subjects.
* Positive urine pregnancy test at screening (performed on all females).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-09; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, MD, Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc., Sainte-Foy, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Amoxicillin Clavulanic Acid (Test) First: Amoxicillin-Clavulanic Acid 400/57 mg chewable tablet (test) dosed in first period followed by Augmentin® 400/57 mg chewable tablet (reference) dosed in second period
- Augmentin® (Reference) First: Augmentin® 400/57 mg chewable tablet (reference) dosed in first period followed by Amoxicillin-Clavulanic Acid 400/57 mg chewable tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Amoxicillin Clavulanic Acid (Test) First | Augmentin® (Reference) First
Started | 24 | 28
Completed | 23 | 28
Not Completed | 1 | 0
Not completed — Difficulty with vein | 1 | 0
Period: Second Intervention
Arm/Group | Amoxicillin Clavulanic Acid (Test) First | Augmentin® (Reference) First
Started | 23 | 28
Completed | 22 | 28
Not Completed | 1 | 0
Not completed — Difficulty with vein | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Amoxicillin Clavulanic Acid (Test) First | Augmentin® (Reference) First | Total
Number analyzed (Participants) | 24 | 28 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 28 | 52
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 8 | 10 | 18
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 23 | 28 | 51
  Black | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 24 | 28 | 52

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration) - Amoxicillin
Description: Bioequivalence based on Cmax
Time Frame: Blood samples were collected over 10 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Amoxicillin Clavulanic Acid: Amoxicillin-Clavulanic Acid 400/57 mg chewable tablet (test) dosed in either period
- Augmentin®: Augmentin® 400/57 mg chewable tablet (reference) dosed in either period
Arm/Group | Amoxicillin Clavulanic Acid | Augmentin®
Number analyzed (Participants) | 50 | 50
ng/mL | 7800.48 (2113.68) | 7599.29 (2222.97)
Statistical Analysis 1: Comparison: Amoxicillin Clavulanic Acid vs Augmentin®; Test type: Non-Inferiority or Equivalence — Using GLM procedures in SAS, analysis of variance (ANOVA)was performed on log-transformed AUC0-t, AUC0-inf and Cmax at the significance level of 0.05; Ratio of Least Squares Means = 103.03, 90% CI [98.40 to 107.88] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

2. Primary Outcome: AUC0-inf - [Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)] - Amoxicillin
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples were collected over 10 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Amoxicillin Clavulanic Acid | Augmentin®
Number analyzed (Participants) | 50 | 50
ng*h/mL | 19089.36 (3440.49) | 19395.97 (3670.87)
Statistical Analysis 1: Comparison: Amoxicillin Clavulanic Acid vs Augmentin®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means = 98.43, 90% CI [96.71 to 100.18] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

3. Primary Outcome: AUC0-t [Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)] - Amoxicillin
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples were collected over 10 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Amoxicillin Clavulanic Acid | Augmentin®
Number analyzed (Participants) | 50 | 50
ng*h/mL | 18939.13 (3441.02) | 19263.26 (3640.51)
Statistical Analysis 1: Comparison: Amoxicillin Clavulanic Acid vs Augmentin®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means = 98.29, 90% CI [96.58 to 100.03] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

4. Primary Outcome: Cmax (Maximum Observed Concentration) - Clavulanic Acid
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 10 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Amoxicillin Clavulanic Acid | Augmentin®
Number analyzed (Participants) | 50 | 50
ng/mL | 1483.32 (508.73) | 1449.68 (497.08)
Statistical Analysis 1: Comparison: Amoxicillin Clavulanic Acid vs Augmentin®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means = 103.16, 90% CI [95.33 to 111.64] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

5. Primary Outcome: AUC0-inf [Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)] - Clavulanic Acid
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 10 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Amoxicillin Clavulanic Acid | Augmentin®
Number analyzed (Participants) | 50 | 50
ng*h/mL | 2876.99 (1022.59) | 2833.74 (1031.56)
Statistical Analysis 1: Comparison: Amoxicillin Clavulanic Acid vs Augmentin®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means = 103.79, 90% CI [95.75 to 112.50] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

6. Primary Outcome: AUC0-t [Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)] - Clavulanic Acid
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 10 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Amoxicillin Clavulanic Acid | Augmentin®
Number analyzed (Participants) | 50 | 50
ng*h/mL | 2798.69 (1011.64) | 2749.12 (1018.15)
Statistical Analysis 1: Comparison: Amoxicillin Clavulanic Acid vs Augmentin®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Least Squares Means = 104.26, 90% CI [95.76 to 113.52] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.